CLINICAL TRIAL: NCT05267119
Title: Comparison of Scalp Microbiome of Healthy Women Wearing Hijab and Those Who do Not Wear Hijab
Status: Completed | Type: Observational
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Dr. dr. Sandra Widaty, SpKK (K), Head of Research and Development Division, Department of Dermatology and Venereology, Indonesia University
Other Study IDs: 19-04-0438
Record Dates: First submitted 2022-02-15; First posted 2022-03-04 (Actual); Last update posted 2022-03-04 (Actual); Status verified 2022-02

CONDITIONS: Microbial Colonization; Scalp--Diseases
Keywords: scalp; microbiome; hijab
MeSH Terms: conditions — Communicable Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Skin
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hijab: Women wearing hijab whose scalp sample was taken for microbiome analysis
  Interventions: Procedure: Swab
- No hijab: Women not wearing hijab whose scalp sample was taken for microbiome analysis
  Interventions: Procedure: Swab

INTERVENTIONS:
Procedure: Swab — The scalp was swabbed with five strokes which were performed each in a vertical, horizontal, left diagonal, and right diagonal direction. The swab was moved back and forth for 10 times

SUMMARY:
An observational study was performed on 48 women wearing hijab and 48 women not wearing hijab to compare the scalp microbiome.

DETAILED DESCRIPTION:
The scalp sample of all subjects was taken to be analyzed for its microbial diversity. The samples were processed with Next-Generation Sequencer and analyzed with bioinformatics analysis.

The primary outcome was the characteristics of scalp microbiome

ELIGIBILITY:
Inclusion Criteria:

* Healthy women
* Aged 18 years old or older who had not undergone menopause
* Consenting to the study

Exclusion Criteria:

* Scalp and hair diseases (e.g. alopecia, trichotillomania, scalp infection, malignancy)
* Systemic diseases (diabetes mellitus, liver diseases, renal diseases, autoimmune diseases)
* Use of topical and oral antifungal agents
* Use of cytostatic agents
* Use of topical and oral antibiotics
* Use of topical and oral vitamin D
* Use of chemical products on hair (e.g. bleaching, permanent blow, hair coloring, hair straightener)
* Pregnancy
* Lactating
* Hypersensitivity towards basic ingredients of shampoo (e.g. synthetic detergent, conditioner, thickening agent).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy women aged 18 years old or older who had not undergone menopause
Sampling Method: Non-Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-11-09 (Actual); Study Completion 2020-11-09 (Actual)

PRIMARY OUTCOMES:
Alpha diversity and beta diversity of scalp microbiome | Up to 2 years
  The alpha and beta diversity of scalp microbiome which is generated by bioinformatics analysis from the sample processed with Next-Generation Sequencing

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Universitas Indonesia, Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No